CLINICAL TRIAL: NCT00212056
Title: Japan-Working Groups of Acute Myocardial Infarction for the Reduction of Necrotic Damage by ANP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Collaborators: Japan Cardiovascular Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSSCJ-1; UMIN_ID:C000000088
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Atrial natriuretic peptide; Data mining; Randomized clinical trial; SNPs

ARMS (2):
- ANP (Active Comparator)
  Interventions: Drug: ANP(hANP)
- Control (Placebo Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: ANP(hANP) — 0∙025 μg/kg per min for 3 days(intravenous)
  Arms: ANP
Drug: Control — placebo
  Arms: Control

SUMMARY:
To evaluate whether ANP as an adjunctive therapy for AMI reduces myocardial infarct size and improves regional wall motion.

DETAILED DESCRIPTION:
The benefits of percutaneous coronary intervention (PCI) in acute myocardial infarction (AMI) are limited by reperfusion injury. In animal models, atrial natriuretic peptide (ANP) reduces infarct size, so the Japan-Working groups of acute myocardial Infarction for the reduction of Necrotic Damage by ANP(J-WINDANP) designed a prospective, randomized, multicenter study, to evaluate whether ANP as an adjunctive therapy for AMI reduces myocardial infarct size and improves regional wall motion.

Twenty hospitals in Japan will participate in the J-WIND-ANP study. Patients with AMI who are candidates for PCI are randomly allocated to receive either intravenous ANP or placebo administration. The primary end-points are (1) estimated infarct size (Σcreatine kinase and troponin T) and (2) left ventricular function (left ventriculograms). Single nucleotide polymorphisms (SNPs) that may be associated with the function of ANP and susceptibility of AMI will be examined. Furthermore, a data mining method will be used to design the optimal combinational therapy for post-MI patients.

J-WIND-ANP will provide important data on the effects of ANP as an adjunct to PCI for AMI and the SNPs information will open the field of tailor-made therapy. The optimal therapeutic drug combination will also be determined for post-MI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-79 years
2. Chest pain of more than 30 min
3. 0.1 mV ST-segment elevation in 2 contiguous ECG leads
4. Admission to hospital within 12 h of symptom onset
5. First episode of AMI
6. Candidates for PCI

Exclusion Criteria:

1. History of old myocardial infarction
2. Left main coronary artery stenosis
3. Severe liver and/or kidney dysfunction
4. Suspected aortic dissection
5. History of coronary artery bypass graft
6. History of allergic response to drugs
7. Severe hypovolemia
8. Right ventricular infarction

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2001-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
estimated infarct size | 72hrs
left ventricular function (left ventricular ejection fraction and end-diastolic volume) and regional wall motion | 2-8weeks and 6-12months

SECONDARY OUTCOMES:
survival rate | 2.7years (median follow-up)
cardiovascular events (ie, cardiac death, nonfatal re-infarction, re-hospitalization because of cardiac disease, revascularization) | 2.7years (median follow-up)
reperfusion injury (ie, malignant ventricular arrhythmia during reperfusion periods, re-elevation of ST-segment, worsening of chest pain) | 24hrs
the association of SNPs of ANP-related genes with response to ANP treatment | 2.7years (median follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Masafumi Kitakaze, MD, PhD, Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Background] Minamino T, Jiyoong K, Asakura M, Shintani Y, Asanuma H, Kitakaze M; J-WIND Investigators. Rationale and design of a large-scale trial using nicorandil as an adjunct to percutaneous coronary intervention for ST-segment elevation acute myocardial infarction: Japan-Working groups of acute myocardial infarction for the reduction of Necrotic Damage by a K-ATP channel opener (J-WIND-KATP). Circ J. 2004 Feb;68(2):101-6. doi: 10.1253/circj.68.101. PMID 14745142